CLINICAL TRIAL: NCT04715399
Title: University of Pennsylvania Centralized Observational Research Repository on Neurodegenerative Disease (UNICORN)
Brief Title: UPenn Observational Research Repository on Neurodegenerative Disease
Acronym: UNICORN
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH); United States Department of Defense (U.S. Federal Agency); National Institute on Aging (NIA) (NIH); Alzheimer's Association (Other)
Responsible Party: Sponsor
Other Study IDs: 842873; R01AG054519 (NIH); P01AG066597 (NIH)
Record Dates: First submitted 2021-01-11; First posted 2021-01-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Frontotemporal Degeneration(FTD); Primary Progressive Aphasia(PPA); Familial Frontotemporal Lobar Degeneration (fFTLD); Amyotrophic Lateral Sclerosis(ALS); Lewy Body Disease(LBD); Progressive Supranuclear Palsy(PSP); Corticobasal Syndrome(CBS); Posterior Cortical Atrophy(PCA); Alzheimer's Disease(AD)
MeSH Terms: conditions — Aphasia, Primary Progressive; Amyotrophic Lateral Sclerosis; Lewy Body Disease; Supranuclear Palsy, Progressive; Corticobasal Degeneration; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples, cerebrospinal fluid (CSF) samples, and saliva or buccal samples may be taken and stored for DNA, RNA and protein extraction and analysis at the University of Pennsylvania and/or research collaborators elsewhere.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cross-sectional
  Interventions: Other: No intervention
- Longitudinal
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The aim of this study is to create a repository of both cross-sectional and longitudinal data, including cognitive, linguistic, imaging and biofluid biological specimens, for neurodegenerative disease research and treatment.

DETAILED DESCRIPTION:
The Principal Investigator (PI) at the University of Pennsylvania seeks to better understand neurodegenerative diseases and is continually expanding research efforts and collaborations regarding the factors which may contribute to these illnesses. Investigators seek to better understand the basis of neurodegenerative conditions by creating a multimodal repository, including: clinical data such as demographic characteristics, vital signs and motor scales; cognitive and speech data; neuroimaging data; and biological specimens with associated biofluid biomarkers and genetic data. Investigators pursue acquiring these data from neurodegenerative disease patients, people at risk for neurodegenerative disease due to a family history, and unaffected adults. Targeted conditions include frontotemporal degeneration (FTD), primary progressive aphasia PPA), amyotrophic lateral sclerosis (ALS), progressive supranuclear palsy (PSP), corticobasal syndrome (CBS), familial frontotemporal lobar degeneration (fFTLD), non-amnestic variants of Alzheimer's disease including logopenic progressive aphasia and posterior cortical atrophy, and Lewy body disease. This study aims to collect clinical and cognitive data, imaging data, and biospecimen samples from people whose background can inform research and treatment for neurodegenerative diseases, and make these samples and data available to qualified researchers at the University of Pennsylvania and collaborating academic centers and industry partners.

ELIGIBILITY:
Inclusion Criteria:

This protocol will include 3 groups of people:

1. People with a clinical diagnosis of a neurodegenerative disease. such as frontotemporal degeneration(FTD), primary progressive aphasia(PPA), Lewy body disease(LBD), amyotrophic lateral sclerosis(ALS), progressive supranuclear palsy(PSP), corticobasal syndrome(CBS), posterior cortical atrophy(PCA), Alzheimer's disease(AD), Parkinson's disease(PD)
2. People with a family history of neurodegenerative disease who may or may not be symptomatic, and may or may not be mutation carriers such as familial frontotemporal lobar degeneration (fFTLD) or familial ALS,
3. People with no known neurological disease who will provide control data.

Exclusion Criteria:

* Anyone who is under the age of 18.
* Anyone with a condition or in a situation which, in the Investigator's opinion, could confound the study findings or may interfere significantly with a person's participation, including but not limited to neurological, psychological and other medical conditions (such as cardiac, neurosurgical, infectious conditions).
* Individual participants may be excluded from some, but not all, study procedures for safety reasons when they have a contraindication or at the discretion of the Investigator. For example, persons with metal implants which are not MRI-safe will not be able to take part in imaging, and those on blood thinning medications may not be able to take part in lumbar puncture.
* Pregnant women; if a woman becomes pregnant during the study, research activities that may increase risk to the patient and the unborn fetus will be stopped until the end of pregnancy, at which point participation can be resumed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To better understand neurodegenerative diseases, the investigators will include people living with these illnesses, people at risk of developing these illnesses, and people without neurodegenerative disease who wish to contribute to science as controls.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-05-29 (Actual); Primary Completion 2070-05-30 (Estimated); Study Completion 2070-05-30 (Estimated)

PRIMARY OUTCOMES:
Status of progression - changes in neuropsychological tests. | This is a natural history study-participants are followed from date of enrollment until death, withdraw, or funding is no longer available, or until 600 months have passed.
  The changes of neuropsychological tests (well known cognitive measures such as: Naming test, CVLT, MoCA, Oral Trails, etc.) in neurodegenerative diseases over time.

SECONDARY OUTCOMES:
Status of progression - changes in language processing. | This is a natural history study-participants are followed from date of enrollment until death, withdraw, or funding is no longer available, or until 600 months have passed.
  The effect of changes in language processing (e.g. effortful speech, lexical-semantic representations) as categorized by impaired speech fluency, motor speech deficits and semantic memory deficits in neurodegenerative diseases over time.
Status of progression - changes in social disinhibition. | This is a natural history study-participants are followed from date of enrollment until death, withdraw, or funding is no longer available, or until 600 months have passed.
  The effect of changes in social behavioral testing, which categorized by rule violation (social disinhibition) progression in neurodegenerative diseases over time.
Status of progression - changes in biofluids. | This is a natural history study-participants are followed from date of enrollment until death, withdraw, or funding is no longer available, or until 600 months have passed.
  The change of disease status as categorized by biomarkers in biofluids in neurodegenerative diseases over time.
Status of progression -changes in Neuroimaging | This is a natural history study-participants are followed from date of enrollment until death, withdraw, or funding is no longer available, or until 600 months have passed.
  The progressive changes of images in multimodal neuroimaging techniques in neurodegenerative diseases over time.

CONTACTS AND LOCATIONS:
Overall Officials: David Irwin, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Information about study participants will be kept confidential and managed according to the requirements of the Health Insurance Portability and Accountability Act of 1996 (HIPAA). Only deidentified data will be shared. We will not share individual participant identifiable data with other researchers outside of the institution, unless the participant allows us to by signing a separate data release form.